CLINICAL TRIAL: NCT05872568
Title: Efficacy and Safety of Enteric-Coated Mycophenolate Sodium (EC-MPS) in de Novo Kidney Transplant Recipients：A Large, Multiple-Center Prospective Study
Brief Title: Efficacy and Safety of Enteric-Coated Mycophenolate Sodium (EC-MPS) in de Novo Kidney Transplant Recipients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhishui Chen (Other)
Responsible Party: Sponsor-Investigator, Zhishui Chen, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TransMate001
Record Dates: First submitted 2023-03-23; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Kidney Transplant Rejection
Keywords: EC-MPS; Kidney Transplant Rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imitation EC-MPS(Ruiyirong) (Experimental)
  Interventions: Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)
- Original EC-MPS（myfortic） (Active Comparator)
  Interventions: Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS) — The recommended dose range is 360 to 720mg,bid

SUMMARY:
At present, imitation EC-MPS have just come on the market, no clinical studies have confirmed the efficacy and safety of using imitation EC-MPS for immunosuppressive therapy after kidney transplantation. Therefore, there is an urgent need to conduct a multicenter study in China to provide further guidance for the use of imitated mycophenol sodium enteric-coated tablets in kidney transplant patients. Therefore, this study will analyze whether the anti-rejection effect of generic EC-MPS in the treatment of renal transplantation in Chinese population is equivalent to that of the original EC-MPS, in order to provide reference for clinical rational drug use.

DETAILED DESCRIPTION:
Under the premise that tacrolimus is used as basic immunosuppressant, to explore the efficacy and safety of imitation mecophenol sodium enteric-coated tablets (EC-MPS) compared with the original preparation agent (Miv) in Chinese kidney transplant patients.

This study was divided into experimental group and control group. The experimental group was imitation mycophenol sodium enteric-coated tablets, and the control group was original mycophenol sodium enteric-coated tablets. Both groups were treated with the triple immunosuppressive regimen of "Mycopherol sodium enteric-coated tablets (EC-MPS) + tacrolimus (TAC) + glucocorticoid" immediately after transplantation for at least 12 months. Tacrolimus, glucocorticoid and antibody induction can be treated according to the clinical routine diagnosis and treatment path, and no specific restrictions were made in this study

ELIGIBILITY:
Inclusion Criteria:

1. Male and female, aged 18-65;
2. Patients with end-stage renal disease who received live/cadaveric kidney transplantation for the first time;
3. After kidney transplantation, patients were subjected to a routine triple immunosuppressive regimen, namely "mecophenol sodium enteric-coated tablets (EC-MPS) + tacrolimus (TAC) + glucocorticoid" regimen;
4. The patients signed informed consent, were able to follow up regularly and fully collect information related to this study.

Exclusion Criteria:

1. Multi-organ recipients, such as those with heart, lung, liver and other organ transplants;
2. ABO incompatible kidney transplant recipients;
3. HLA antibodies or past/current population reactive antibody level (PRA) > 25% were preexisting in the recipient before renal transplantation;
4. Allergic to EC-MPS or preparation components (hypersensitivity);
5. Women with fertility potential who are pregnant, lactating or planning to become pregnant;
6. Severe/uncontrolled concomitant infections or other serious medical problems;
7. Active bacterial, viral or fungal infections;
8. Neutropenia (ANC<1.3×103/µL)
9. Patients judged by the investigator to be unsuitable for inclusion in this study for other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute rejection | 6 months after renal transplantation
Incidence of acute rejection | 12 months after renal transplantation

SECONDARY OUTCOMES:
Incidence of gastrointestinal reactions | 12 months after renal transplantation

OTHER OUTCOMES:
Graft survival rate | 12 months after renal transplantation
Patients survival rate | 12 months after renal transplantation
adverse event rate | 12 months after renal transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Zhishui Chen, Dr., Principal Investigator — Tongji Hospital Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No